CLINICAL TRIAL: NCT01425801
Title: A Phase IIa, Randomised, Single Dose, Double-blind, Double-dummy, 6 Way Complete Cross-over, Placebo Controlled Clinical Trial to Assess the Efficacy, Safety and Tolerability of 4 Doses of LAS100977 QD Compared to Placebo and an Active Comparator in Patients With Persistent Asthma.
Brief Title: Single Dose Study to Assess Efficacy, Safety and Tolerability of LAS100977 in Asthmatic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M/100977/202
Record Dates: First submitted 2011-08-29; First posted 2011-08-30 (Estimated); Results first posted 2018-01-26 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- LAS100977 0.625 μg (Experimental): Single-dose LAS100977 0.625 μg, during double-blind treatment period
  Interventions: Drug: LAS100977 0.625 μg; Drug: Salbutamol placebo
- LAS100977 1.25 μg (Experimental): Single-dose LAS100977 1.25 μg, during double-blind treatment period
  Interventions: Drug: LAS100977 1.25 μg; Drug: Salbutamol placebo
- LAS100977 2.5 μg (Experimental): Single-dose LAS100977 2.5 μg, during double-blind treatment period
  Interventions: Drug: LAS100977 2.5 μg; Drug: Salbutamol placebo
- Salbutamol (Active Comparator): Single-dose salbutamol 400 μg, during double-blind treatment period
  Interventions: Drug: Salbutamol 400 μg; Drug: LAS100977 placebo
- Placebo (Placebo Comparator): Placebo to LAS100977, and placebo to salbutamol
  Interventions: Drug: Salbutamol placebo; Drug: LAS100977 placebo
- LAS100977 0.313 μg (Experimental): Single-dose LAS100977 0.313 μg, during double-blind treatment period
  Interventions: Drug: LAS100977 0.313 μg; Drug: Salbutamol placebo

INTERVENTIONS:
Drug: LAS100977 0.313 μg — Dry powder inhalation, once-daily, single-dose
  Arms: LAS100977 0.313 μg
Drug: LAS100977 0.625 μg — Dry powder inhalation, once-daily, single-dose
  Arms: LAS100977 0.625 μg
Drug: LAS100977 1.25 μg — Dry powder inhalation, once-daily, single-dose
  Arms: LAS100977 1.25 μg
Drug: LAS100977 2.5 μg — Dry powder inhalation, once-daily, single-dose
  Arms: LAS100977 2.5 μg
Drug: Salbutamol 400 μg — Pressurized inhalation suspension, once-daily, single-dose
  Arms: Salbutamol
Drug: Salbutamol placebo — Pressurized inhalation, once-daily
  Arms: LAS100977 0.313 μg; LAS100977 0.625 μg; LAS100977 1.25 μg; LAS100977 2.5 μg; Placebo
Drug: LAS100977 placebo — Dry powder inhalation, once-daily
  Arms: Placebo; Salbutamol

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamics of single doses of inhaled LAS100977 QD in patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female patients aged 18-70 years (both included).
2. Clinical diagnosis of persistent asthma (according to GINA guidelines 2009 update) for at least 6 months prior to screening.
3. Screening FEV1 value of 60% < FEV1 ≤ 85% of the predicted normal value.
4. FEV1 reversibility ≥ 12% and an absolute increase of at least 200 ml over baseline value after inhalation of 400µg (four inhalations) of salbutamol.
5. Pre-dose FEV1 value of first treatment period within the range of ± 20% of the FEV1 measured at screening prior to salbutamol inhalation.
6. Patients on a stable dose and regimen

Exclusion Criteria:

1. Current smokers, former smokers within the last 6 months, or ex-smokers with a history of more than 10 pack-years.
2. Patients diagnosed with COPD.
3. Recent Respiratory tract infections within 6 weeks before Screening Visit.
4. Intubation (ever) or hospitalization for longer than 24 hours for the management of an asthma exacerbation within the preceding 6 weeks of the screening visit.
5. Clinically significant respiratory conditions.
6. Clinically significant cardiovascular conditions.
7. Patients unable to properly use a dry powder or pMDI inhaler device or unable to perform acceptable spirometry.
8. Clinically relevant abnormalities laboratory, ECG parameters or physical examination results at the screening evaluation that in the investigator's opinion, preclude study participation.
9. Patients who intend to use any concomitant medication not permitted by this protocol or who have not undergone the required washout period for a particular prohibited medication.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2012-02-01 (Actual); Study Completion 2012-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Astbury, PhD, Study Director — AstraZeneca
Locations (9):
- Germany (7):
  - Almirall Investigational Sites#6, Berlin
  - Almirall Investigational Sites#4, Berlin
  - Almirall Investigational Sites#1, Berlin
  - Almirall Investigational Sites#3, Frankfurt
  - Almirall Investigational Sites#2, Großhansdorf
  - Almirall Investigational Sites#8, Hamburg
  - Almirall Investigational Sites#5, Wiesbaden
- United Kingdom (2):
  - Almirall Investigational Sites#2, London
  - Almirall Investigational Sites#1, Manchester

REFERENCES:
- [Derived] Singh D, Pujol H, Ribera A, Seoane B, Massana E, Astbury C, Ruiz S, de Miquel G. A dose-ranging study of the bronchodilator effects of abediterol (LAS100977), a long-acting beta2-adrenergic agonist, in asthma; a Phase II, randomized study. BMC Pulm Med. 2014 Nov 14;14:176. doi: 10.1186/1471-2466-14-176. PMID 25398689
- See also: Synopsis-M-100977-202 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3968&filename=Synopsis-M-100977-202-Final.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 10 sites in Germany and United Kingdom, 9 of which randomized patients
Pre-assignment Details: Screening took place 12-16 days before randomization. After screening, eligible patients entered a run-in period to assess clinical stability. A total of 115 patients were screened; 62 patients were assessed as eligible and randomized; 53 were not randomized due to screening failure (primarily non-fulfillment of inclusion/exclusion criteria)
Groups:
- Sequence A: Salbutamol 400 μg - LAS100977 0.313 μg - Placebo - LAS100977 0.625 μg - LAS100977 2.5 μg - LAS100977 1.25 μg
- Sequence B: LAS100977 0.313 μg - LAS100977 0.625 μg - Salbutamol 400 μg - LAS100977 1.25 μg - Placebo - LAS100977 2.5 μg
- Sequence C: LAS100977 0.625 μg - LAS100977 1.25 μg - LAS100977 0.313 μg - LAS100977 2.5 μg - Salbutamol 400 μg - Placebo
- Sequence D: LAS100977 1.25 μg - LAS100977 2.5 μg - LAS100977 0.625 μg - Placebo - LAS100977 0.313 μg - Salbutamol 400 μg
- Sequence E: LAS100977 2.5 μg - Placebo - LAS100977 1.25 μg - Salbutamol 400 μg - LAS100977 0.625 μg - LAS100977 0.313 μg
- Sequence F: Placebo - Salbutamol 400 μg - LAS100977 2.5 μg - LAS100977 0.313 μg - LAS100977 1.25 μg - LAS100977 0.625 μg
Period: Period 1
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 9 | 9 | 12 | 13 | 10
Completed | 9 | 9 | 9 | 12 | 12 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 9 | 9 | 12 | 12 | 10
Completed | 9 | 9 | 9 | 12 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 3
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 9 | 9 | 12 | 11 | 10
Completed | 9 | 9 | 8 | 12 | 11 | 10
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Stability criteria not fullfilled | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 9 | 8 | 12 | 11 | 10
Completed | 9 | 9 | 7 | 12 | 11 | 10
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Not able to maintain visit schedule | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 9 | 7 | 12 | 11 | 10
Completed | 9 | 9 | 7 | 12 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6
Arm/Group | Sequence A | Sequence B | Sequence C | Sequence D | Sequence E | Sequence F
Started | 9 | 9 | 7 | 12 | 11 | 10
Completed | 9 | 9 | 7 | 12 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Population: Safety population defined as all patients who were randomized and received at least one dose of investigational medicinal product
Arm/Group | Overall Population
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Peak Forced Expiratory Volume in One Second (FEV1)
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). The peak was computed as the highest value observed for each patient during the 4-hour period immediately after the investigational medicinal product administered in the morning. At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 were selected.
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h post-dose
Population: ITT population defined as patients who took at least one dose of investigational medicinal product and had at least a baseline and one post-dose value of FEV1 from at least one treatment period
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Placebo: Dry powder administered via the Genuair® inhaler or pressurised inhalation suspension administered via Ventolin Evohaler®
- LAS100977 0.313 μg: Dry powder administered via the Genuair® inhaler
- LAS100977 0.625 μg; LAS100977 1.25 μg; LAS100977 2.5 μg: Dry powder for inhalation administered via Genuair®
- Salbutamol 400 μg: Pressurised inhalation suspension administered via Ventolin Evohaler®
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters | 0.202 (0.045) | 0.477 (0.045) | 0.524 (0.045) | 0.573 (0.045) | 0.608 (0.045) | 0.555 (0.045)
Statistical Analysis 1: Comparison: Placebo vs LAS100977 2.5 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Sequence, treatment and period as fixed effect factors, patient within sequence as random effect and baseline peak FEV1 at each period as a covariate; Least Squares Mean DIfference = 0.405, 95% CI 2-sided [0.353 to 0.458], Standard Error of Mean 0.027
Statistical Analysis 2: Comparison: Placebo vs LAS100977 1.25 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.371, 95% CI 2-sided [0.318 to 0.424], Standard Error of Mean 0.027
Statistical Analysis 3: Comparison: Placebo vs LAS100977 0.625 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.322, 95% CI 2-sided [0.269 to 0.375], Standard Error of Mean 0.027
Statistical Analysis 4: Comparison: Placebo vs LAS100977 0.313 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Least Squares Mean Difference = 0.274, 95% CI 2-sided [0.221 to 0.327], Standard Error of Mean 0.027

2. Secondary Outcome: Percentage Change From Baseline in Peak Forced Expiratory Volume in One Second (FEV1)
Description: as for outcome 1
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Percent change | 7.555 (1.655) | 18.282 (1.651) | 20.212 (1.651) | 21.809 (1.651) | 23.077 (1.650) | 21.374 (1.658)

3. Secondary Outcome: Peak Forced Expiratory Volume in One Second (FEV1)
Description: The peak was computed as the highest value observed for each patient during the 4-hour period immediately after the investigational medicinal product administered in the morning on Day 1. At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 were selected.
Time Frame: +15 min, +30 min, +1 h, +2 h, +3 h, +4 h post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters | 2.855 (0.045) | 3.129 (0.045) | 3.177 (0.045) | 3.225 (0.045) | 3.260 (0.045) | 3.207 (0.045)

4. Secondary Outcome: Time to Peak Forced Expiratory Volume in One Second (FEV1)
Description: The peak was computed as the highest value observed for each patient during the 4-hour period immediately after the investigational medicinal product administered in the morning. At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 were selected.
Time Frame: +15 min, +30 min, +1 h, +2 h, +3 h, +4 h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Hours | 2.3 (1.3) | 2.6 (1.3) | 3.0 (1.1) | 3.1 (0.9) | 3.0 (1.1) | 1.1 (0.8)

5. Secondary Outcome: Change From Baseline to Trough Forced Expiratory Volume in One Second (FEV1)
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). Trough at Day 2 was computed as the average of the two values measured at 23 and 24 hours after administration of the morning dose of investigational medicinal product on Day 1. At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected.
Time Frame: Baseline and +23 h and +24 h post-dose
Population: Patients in the ITT population with available data at the timepoints of interest. ITT population defined as patients who took at least one dose of investigational medicinal product and had at least a baseline and one post-dose value of FEV1 from at least one treatment period
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
Liters | -0.054 (0.039) | 0.166 (0.039) | 0.205 (0.039) | 0.278 (0.039) | 0.346 (0.039) | -0.076 (0.039)

6. Secondary Outcome: Change From Baseline in Normalized Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC) 0-24h at Day 1
Description: FEV1 was normalized to baseline. Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected.
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h and +24 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 57 | 59 | 60 | 60 | 59 | 53
Liters | 0.007 (0.039) | 0.282 (0.039) | 0.321 (0.038) | 0.390 (0.038) | 0.446 (0.039) | 0.100 (0.039)

7. Secondary Outcome: Absolute Values of Forced Expiratory Volume (FEV1) at Each Timepoint
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected.
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h, +24 h, and +36 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters
  0.25 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 57
  0.25 hr | 2.696 (0.030) | 2.863 (0.030) | 2.886 (0.030) | 2.934 (0.030) | 3.007 (0.030) | 3.106 (0.030)
  1 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  1 hr | 2.719 (0.037) | 3.000 (0.037) | 3.025 (0.037) | 3.098 (0.037) | 3.133 (0.037) | 3.147 (0.037)
  2 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  2 hr | 2.746 (0.039) | 3.034 (0.038) | 3.081 (0.038) | 3.136 (0.038) | 3.188 (0.039) | 3.123 (0.039)
  3 hr: number analyzed (Participants) | 59 | 60 | 60 | 59 | 61 | 58
  3 hr | 2.771 (0.041) | 3.069 (0.041) | 3.102 (0.041) | 3.190 (0.041) | 3.196 (0.041) | 3.040 (0.041)
  4 hr | 2.774 (0.044) | 3.058 (0.044) | 3.124 (0.044) | 3.167 (0.044) | 3.211 (0.044) | 2.937 (0.044)
  6 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 61 | 58
  6 hr | 2.722 (0.038) | 3.008 (0.038) | 3.087 (0.038) | 3.157 (0.038) | 3.194 (0.038) | 2.812 (0.038)
  8 hr: number analyzed (Participants) | 57 | 60 | 60 | 60 | 61 | 58
  8 hr | 2.715 (0.040) | 3.033 (0.039) | 3.062 (0.039) | 3.139 (0.039) | 3.180 (0.039) | 2.772 (0.039)
  12 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 56
  12 hr | 2.659 (0.044) | 2.943 (0.043) | 2.980 (0.043) | 3.035 (0.043) | 3.111 (0.043) | 2.669 (0.044)
  14 hr: number analyzed (Participants) | 58 | 59 | 60 | 60 | 59 | 53
  14 hr | 2.597 (0.042) | 2.903 (0.041) | 2.941 (0.041) | 3.018 (0.041) | 3.094 (0.042) | 2.683 (0.043)
  23 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  23 hr | 2.588 (0.040) | 2.804 (0.039) | 2.836 (0.040) | 2.923 (0.040) | 2.985 (0.040) | 2.562 (0.040)
  24 hr: number analyzed (Participants) | 58 | 60 | 59 | 59 | 60 | 57
  24 hr | 2.618 (0.040) | 2.840 (0.039) | 2.890 (0.040) | 2.948 (0.040) | 3.019 (0.040) | 2.605 (0.040)
  36 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  36 hr | 2.689 (0.042) | 2.823 (0.041) | 2.798 (0.041) | 2.892 (0.041) | 2.929 (0.041) | 2.690 (0.041)
  0.5 hr | 2.723 (0.034) | 2.956 (0.033) | 2.972 (0.033) | 3.033 (0.033) | 3.089 (0.033) | 3.142 (0.034)

8. Secondary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1) at Each Timepoint
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected. The number of participants analyzed differed between timepoints - the number of participants analyzed at 0.25 h is shown.
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h, +24 h, and +36 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters
  0.25 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 57
  0.25 hr | 0.048 (0.030) | 0.214 (0.030) | 0.237 (0.030) | 0.285 (0.030) | 0.358 (0.030) | 0.457 (0.030)
  0.5 hr | 0.071 (0.034) | 0.304 (0.033) | 0.319 (0.033) | 0.381 (0.033) | 0.437 (0.033) | 0.490 (0.034)
  1 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  1 hr | 0.067 (0.037) | 0.348 (0.037) | 0.373 (0.037) | 0.446 (0.037) | 0.481 (0.037) | 0.495 (0.037)
  2 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  2 hr | 0.094 (0.039) | 0.382 (0.038) | 0.429 (0.038) | 0.484 (0.038) | 0.536 (0.039) | 0.471 (0.039)
  3 hr: number analyzed (Participants) | 59 | 60 | 60 | 59 | 61 | 58
  3 hr | 0.119 (0.041) | 0.416 (0.041) | 0.450 (0.041) | 0.537 (0.041) | 0.543 (0.041) | 0.388 (0.041)
  4 hr | 0.121 (0.044) | 0.406 (0.044) | 0.471 (0.044) | 0.515 (0.044) | 0.558 (0.044) | 0.284 (0.044)
  6 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 61 | 58
  6 hr | 0.067 (0.038) | 0.353 (0.038) | 0.432 (0.038) | 0.501 (0.038) | 0.539 (0.038) | 0.157 (0.038)
  8 hr: number analyzed (Participants) | 57 | 60 | 60 | 60 | 61 | 58
  8 hr | 0.056 (0.040) | 0.374 (0.039) | 0.403 (0.039) | 0.480 (0.039) | 0.521 (0.039) | 0.113 (0.039)
  12 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 56
  12 hr | 0.005 (0.044) | 0.288 (0.043) | 0.326 (0.043) | 0.380 (0.043) | 0.456 (0.043) | 0.014 (0.044)
  14 hr: number analyzed (Participants) | 58 | 59 | 60 | 60 | 59 | 53
  14 hr | -0.053 (0.042) | 0.253 (0.041) | 0.291 (0.041) | 0.367 (0.041) | 0.443 (0.042) | 0.032 (0.043)
  23 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  23 hr | -0.067 (0.040) | 0.148 (0.039) | 0.181 (0.040) | 0.268 (0.040) | 0.330 (0.040) | -0.093 (0.040)
  24 hr: number analyzed (Participants) | 58 | 60 | 59 | 59 | 60 | 57
  24 hr | -0.040 (0.040) | 0.183 (0.039) | 0.233 (0.040) | 0.291 (0.040) | 0.362 (0.040) | -0.052 (0.040)
  36 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  36 hr | 0.035 (0.042) | 0.169 (0.041) | 0.144 (0.041) | 0.238 (0.041) | 0.275 (0.041) | 0.036 (0.041)

9. Secondary Outcome: Percentage Change From Baseline in Forced Expiratory Volume (FEV1) at Each Timepoint
Description: as for outcome 8
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h, +24 h, and +36 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Percent change
  0.25 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 57
  0.25 hr | 1.519 (1.090) | 8.325 (1.084) | 8.846 (1.084) | 10.789 (1.084) | 13.511 (1.081) | 17.744 (1.098)
  0.5 hr | 2.449 (1.205) | 11.757 (1.199) | 12.006 (1.199) | 14.362 (1.199) | 16.715 (1.196) | 18.806 (12.209)
  1 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  1 hr | 2.407 (1.356) | 13.452 (1.350) | 14.307 (1.350) | 16.927 (1.350) | 18.336 (1.352) | 19.085 (1.360)
  2 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  2 hr | 3.520 (1.434) | 14.741 (1.427) | 16.371 (1.428) | 18.509 (1.428) | 20.226 (1.430) | 17.755 (1.438)
  3 hr: number analyzed (Participants) | 59 | 60 | 60 | 59 | 61 | 58
  3 hr | 4.435 (1.479) | 15.965 (1.472) | 17.190 (1.472) | 20.357 (1.477) | 20.550 (1.470) | 14.537 (1.484)
  4 hr | 4.288 (1.596) | 15.400 (1.589) | 17.960 (1.590) | 19.454 (1.590) | 21.155 (1.587) | 10.608 (1.600)
  6 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 61 | 58
  6 hr | 2.682 (1.439) | 13.661 (1.424) | 16.490 (1.425) | 19.080 (1.425) | 20.612 (1.421) | 5.796 (1.438)
  8 hr: number analyzed (Participants) | 57 | 60 | 60 | 60 | 61 | 58
  8 hr | 2.752 (1.505) | 14.118 (1.482) | 15.128 (1.482) | 18.199 (1.482) | 19.733 (1.478) | 4.493 (1.497)
  12 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 56
  12 hr | 0.402 (1.627) | 10.847 (1.614) | 12.388 (1.614) | 14.251 (1.614) | 17.170 (1.616) | 0.997 (1.639)
  14 hr: number analyzed (Participants) | 58 | 59 | 60 | 60 | 59 | 53
  14 hr | -1.903 (1.559) | 9.427 (1.551) | 11.008 (1.544) | 11.771 (1.544) | 16.716 (1.555) | 1.892 (1.594)
  23 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  23 hr | -2.117 (1.464) | 5.451 (1.444) | 6.955 (1.445) | 9.893 (1.445) | 12.375 (1.449) | -3.649 (1.464)
  24 hr: number analyzed (Participants) | 58 | 60 | 59 | 59 | 60 | 57
  24 hr | -0.611 (1.473) | 7.084 (1.453) | 8.918 (1.461) | 10.975 (1.461) | 13.716 (1.458) | -1.736 (1.482)
  36 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  36 hr | 1.904 (1.574) | 6.396 (1.554) | 5.589 (1.555) | 8.742 (1.555) | 10.370 (1.558) | 2.098 (1.572)

10. Secondary Outcome: Change From Baseline in Peak Forced Vital Capacity (FVC)
Description: Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). The peak was computed as the highest value observed for each patient during the 4-hour period immediately after the investigational medicinal product administered in the morning. At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected.
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h post-dose
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters | 0.222 (0.034) | 0.317 (0.034) | 0.329 (0.034) | 0.361 (0.034) | 0.380 (0.034) | 0.361 (0.034)

11. Secondary Outcome: Peak Forced Vital Capacity (FVC)
Description: The peak was computed as the highest value observed for each patient during the 4-hour period immediately after the investigational medicinal product administered in the morning. At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected.
Time Frame: +15 min, +30 min, +1 h, +2 h, +3 h, +4 h
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters | 4.483 (0.034) | 4.578 (0.034) | 4.590 (0.034) | 4.622 (0.034) | 4.641 (0.034) | 4.622 (0.034)

12. Secondary Outcome: Time to Peak Forced Vital Capacity (FVC)
Description: as for outcome 11
Time Frame: +15 min, +30 min, +1 h, +2 h, +3 h, +4 h
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Hours | 2.1 (1.4) | 1.8 (1.4) | 2.3 (1.4) | 2.1 (1.2) | 2.2 (1.4) | 1.5 (1.2)

13. Secondary Outcome: Change From Baseline to Trough Forced Vital Capacity (FVC)
Description: as for outcome 5
Time Frame: Baseline and +23 h +24 h post-dose
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
Liters | -0.028 (0.035) | 0.094 (0.035) | 0.050 (0.035) | 0.111 (0.035) | 0.120 (0.035) | -0.065 (0.035)

14. Secondary Outcome: Change From Baseline in Normalized Forced Vital Capacity (FVC) Area Under the Curve (AUC)
Description: FVC was normalized to baseline. Baseline was the average of the two values measured just prior to the administration of the dose of investigational medicinal product at Day 1 of each visit (time points -45 min and -15 min). At each time point, three technically adequate lung function measurements were performed by spirometry according to the acceptability and repeatability criteria of the ATS/ERS; the highest values for the FEV1 and FVC were selected.
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h and +24 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 57 | 59 | 60 | 60 | 59 | 53
Liters | 0.017 (0.031) | 0.135 (0.031) | 0.109 (0.030) | 0.169 (0.030) | 0.192 (0.031) | 0.054 (0.031)

15. Secondary Outcome: Absolute Values of Forced Vital Capacity (FVC) at Each Timepoint
Description: as for outcome 8
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h, +24 h, and +36 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters
  0.25h: number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 57
  0.25h | 4.295 (0.030) | 4.420 (0.030) | 4.368 (0.030) | 4.383 (0.030) | 4.417 (0.030) | 4.471 (0.030)
  0.5 hr | 4.320 (0.032) | 4.458 (0.032) | 4.405 (0.032) | 4.438 (0.032) | 4.443 (0.032) | 4.502 (0.032)
  1 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  1 hr | 4.295 (0.034) | 4.442 (0.034) | 4.429 (0.034) | 4.480 (0.034) | 4.498 (0.034) | 4.502 (0.034)
  2 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  2 hr | 4.321 (0.034) | 4.445 (0.034) | 4.444 (0.034) | 4.495 (0.034) | 4.512 (0.034) | 4.477 (0.034)
  3 hr: number analyzed (Participants) | 59 | 60 | 60 | 59 | 61 | 58
  3 hr | 4.352 (0.036) | 4.462 (0.035) | 4.472 (0.035) | 4.505 (0.035) | 4.505 (0.035) | 4.454 (0.036)
  4 hr | 4.316 (0.035) | 4.459 (0.035) | 4.462 (0.035) | 4.463 (0.035) | 4.517 (0.034) | 4.398 (0.035)
  6 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 61 | 58
  6 hr | 4.322 (0.033) | 4.413 (0.033) | 1.411 (0.033) | 4.464 (0.033) | 4.513 (0.033) | 4.360 (0.033)
  8 hr: number analyzed (Participants) | 57 | 60 | 60 | 60 | 61 | 58
  8 hr | 4.325 (0.035) | 4.456 (0.035) | 4.412 (0.035) | 4.487 (0.035) | 4.499 (0.035) | 4.335 (0.035)
  12 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 56
  12 hr | 4.310 (0.036) | 4.409 (0.036) | 4.349 (0.036) | 4.414 (0.036) | 4.453 (0.036) | 4.277 (0.037)
  14 hr: number analyzed (Participants) | 58 | 59 | 60 | 60 | 59 | 53
  14 hr | 4.235 (0.036) | 4.357 (0.036) | 4.360 (0.036) | 4.436 (0.036) | 4.458 (0.036) | 4.269 (0.037)
  23 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  23 hr | 4.244 (0.037) | 4.366 (0.036) | 4.303 (0.036) | 4.375 (0.036) | 4.367 (0.036) | 4.223 (0.037)
  24 hr: number analyzed (Participants) | 58 | 60 | 59 | 59 | 60 | 57
  24 hr | 4.238 (0.038) | 4.359 (0.037) | 4.335 (0.038) | 4.384 (0.038) | 4.410 (0.038) | 4.193 (0.038)
  36 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  36 hr | 4.252 (0.040) | 4.390 (0.039) | 4.280 (0.039) | 4.352 (0.039) | 4.381 (0.039) | 4.284 (0.040)

16. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Each Timepoint
Description: as for outcome 8
Time Frame: Baseline and +15 min, +30 min, +1 h, +2 h, +3 h, +4 h, +6 h, +8 h, +12 h, +14 h, +23 h, +24 h, and +36 h
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 58
Liters
  0.25 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 61 | 57
  0.25 hr | 0.038 (0.030) | 0.162 (0.030) | 0.111 (0.030) | 0.125 (0.030) | 0.159 (0.030) | 0.213 (0.030)
  0.5 hr | 0.059 (0.032) | 0.197 (0.032) | 0.144 (0.032) | 0.177 (0.032) | 0.182 (0.032) | 0.241 (0.032)
  1 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  1 hr | 0.034 (0.034) | 0.182 (0.034) | 0.169 (0.034) | 0.219 (0.034) | 0.237 (0.034) | 0.242 (0.034)
  2 hr: number analyzed (Participants) | 59 | 60 | 60 | 60 | 60 | 58
  2 hr | 0.060 (0.034) | 0.184 (0.034) | 0.183 (0.034) | 0.234 (0.034) | 0.252 (0.034) | 0.217 (0.034)
  3 hr: number analyzed (Participants) | 59 | 60 | 60 | 59 | 61 | 58
  3 hr | 0.089 (0.036) | 0.199 (0.035) | 0.209 (0.035) | 0.241 (0.035) | 0.242 (0.035) | 0.191 (0.036)
  4 hr | 0.055 (0.035) | 0.198 (0.035) | 0.201 (0.035) | 0.202 (0.035) | 0.256 (0.034) | 0.137 (0.035)
  6 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 61 | 58
  6 hr | 0.057 (0.033) | 0.149 (0.033) | 0.147 (0.033) | 0.200 (0.033) | 0.249 (0.033) | 0.096 (0.033)
  8 hr: number analyzed (Participants) | 57 | 60 | 60 | 60 | 61 | 58
  8 hr | 0.054 (0.035) | 0.185 (0.035) | 0.141 (0.035) | 0.216 (0.035) | 0.228 (0.035) | 0.064 (0.035)
  12 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 56
  12 hr | 0.042 (0.036) | 0.141 (0.036) | 0.081 (0.036) | 0.146 (0.036) | 0.185 (0.036) | 0.001 (0.037)
  14 hr: number analyzed (Participants) | 58 | 59 | 60 | 60 | 59 | 53
  14 hr | -0.027 (0.036) | 0.095 (0.036) | 0.097 (0.036) | 0.173 (0.036) | 0.195 (0.036) | 0.006 (0.037)
  23 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  23 hr | -0.022 (0.037) | 0.101 (0.036) | 0.038 (0.036) | 0.110 (0.036) | 0.102 (0.036) | -0.043 (0.037)
  24 hr: number analyzed (Participants) | 58 | 60 | 59 | 59 | 60 | 57
  24 hr | -0.034 (0.038) | 0.086 (0.037) | 0.063 (0.038) | 0.111 (0.038) | 0.137 (0.038) | -0.079 (0.038)
  36 hr: number analyzed (Participants) | 58 | 60 | 60 | 60 | 60 | 58
  36 hr | -0.011 (0.040) | 0.128 (0.039) | 0.018 (0.039) | 0.089 (0.039) | 0.118 (0.039) | 0.022 (0.040)

ADVERSE EVENTS:
Time Frame: Up to 14 (±2) days after last intake of investigational medicinal product
Description: Safety population defined as all randomized patients who took at least 1 dose of investigational medicinal product The total number of patients in the safety population was 62; due to study drop-out and the crossover study design, not all patients received all treatments
Arm/Group | Placebo | LAS100977 0.313 μg | LAS100977 0.625 μg | LAS100977 1.25 μg | LAS100977 2.5 μg | Salbutamol 400 μg
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60 | 0/60 | 0/60 | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 8/59 | 12/60 | 10/60 | 12/60 | 9/61 | 6/62
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | LAS100977 0.313 μg (N=60) | LAS100977 0.625 μg (N=60) | LAS100977 1.25 μg (N=60) | LAS100977 2.5 μg (N=61) | Salbutamol 400 μg (N=62)
Headache (Nervous system disorders) | 7 | 4 | 7 | 8 | 7 | 6
Nasopharyngitis (Infections and infestations) | 1 | 8 | 3 | 4 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and/or presentation whether complete or partial, of any part of the data or results of this trial will be subject to revision and written agreement between the investigator and sponsor